CLINICAL TRIAL: NCT07051967
Title: Post-intensive Care Syndromes in Pregnant Patients With Respiratory Failure and COVID-19 Compared to Non-pregnant Patients With Respiratory Failure and COVID-19
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - Universitaetsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: CovPreg
Record Dates: First submitted 2025-07-03; First posted 2025-07-04 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: COVID-19; Acute Respiratory Distress Syndrome Due to COVID-19; Pregnancy Related
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female pregnant patients with COVID-19 related Acute respiratory distress syndrome: * Pregnancy at the time of initial hospital admission (not necessarily at the time of transfer to Charité - Universitätsmedizin Berlin).
  * Age: 18 years and older
  * Admission to a Charité intensive care unit and follow-up examination by the Post-Intensive-Care-Syndrome (PICS) outpatient clinic of the Department of Anesthesiology and Intensive Care Medicine between March 27, 2020 and May 6, 2024.
  * COVID-19 infection in temporal association with the intensive care unit admission.
  * Intensive care unit admission with lung failure or development of lung failure in the course of intensive care unit treatment.
  * Admission to the intensive care unit with lung failure or development of lung failure during intensive care unit stay
- Female non-pregnant patients with COVID-19 related Acute respiratory distress syndrome: * No pregnancy at the time of admission.
  * Age: 18 years and older
  * Admission to a Charité intensive care unit and follow-up examination by the Post-Intensive-Care-Syndrome (PICS) outpatient clinic of the Department of Anesthesiology and Intensive Care Medicine between March 27, 2020 and May 6, 2024.
  * COVID-19 infection in temporal association with the intensive care unit admission.
  * Intensive care unit admission with lung failure or development of lung failure in the course of intensive care unit treatment.
  * Admission to the intensive care unit with lung failure or development of lung failure during intensive care unit stay

SUMMARY:
The aim of this study is to characterize patients in the Post-Intensive-Care-Syndrome (PICS) outpatient clinic based on routine data and to evaluate their treatment outcome over the course of their treatment. For this purpose, data sets from approx. 40 patients who were treated in the intensive care unit subsequently evaluated in the PICS outpatient clinic between March 27, 2020, and May 6, 2024, will be analyzed.

DETAILED DESCRIPTION:
This is a retrospective comparison of approximately 13 pregnant patients and approximately 27 non-pregnant patients who developed respiratory failure (also known as acute respiratory distress syndrome, or ARDS) due to COVID-19 infection. The analysis is based on routine treatment data from the Post-Intensive Care Syndrome (PICS) outpatient clinic of the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), as well as intensive care treatment data, primarily from the Department of Anesthesiology and Intensive Care Medicine (CCM/CVK). In some cases, additional data were obtained from the Medical Clinic for Nephrology and Internal Intensive Care Medicine (CCM/CVK/CBF), the Medical Clinic specializing in Hepatology and Gastroenterology (CCM/CVK), and the Department of Infectiology, Pulmonology, and Intensive Care Medicine (CCM).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older
* Admission to a Charité intensive care unit and follow-up examination by the Post-Intensive-Care-Syndrome (PICS) outpatient clinic of the Department of Anesthesiology and Intensive Care Medicine between March 27, 2020 and May 6, 2024.
* COVID-19 infection in temporal assocoation with the intensive care unit admission.
* Intensive care unit admission with lung failure or development of lung failure in the course of intensive care unit treatment.
* Admission to the intensive care unit with lung failure or development of lung failure during intensive care unit stay.

Exclusion Criteria:

* Gender: Male
* Diagnosis: Non-COVID or no respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female pregnant and non-pregnant patients who were admitted to a Charité intensive care unit and follow-up examination by the Post-Intensive-Care-Syndrome (PICS) outpatient clinic of the Department of Anesthesiology and Intensive Care Medicine, Charité - Universitaetsmedizin Berlin between March 27, 2020 and May 6, 2024.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Impairment in at least one PICS domain (mobility, cognition, and/or mental health) | 27.03.2020-06.05.2024
  Impairment in at least one PICS domain (mobility, cognition, and/or mental health) after discharge from the ICU, assessed at the time of presentation to the PICS outpatient clinic. The planned PICS outpatient presentation takes place 3 and 6 months (ranging from 1 month to 3 years) after the initial ICU stay.

SECONDARY OUTCOMES:
Catecholamine therapy | 27.03.2020-06.05.2024
  Catecholamine therapy during intensive care unit (ICU) treatment is measured in doses and duration.
Extracorporeal Membrane Oxygenation treatment | 27.03.2020-06.05.2024
  Extracorporeal Membrane Oxygenation treatment in the ICU Yes or No
Need for ventilation during ICU treatment | 27.03.2020-06.05.2024
  Need for ventilation during ICU treatment and, if so, ventilation route (non-invasive and invasive, endotracheal tube and tracheostomy tube) and duration of ventilation
Duration of ventilation during ICU treatment | 27.03.2020-06.05.2024
  Duration of ventilation during ICU treatment is measured in hours
Oxygenation index | 27.03.2020-06.05.2024
  Oxygenation index/Horowitz index is defined as the ratio of the arterial partial pressure of oxygen (PaO₂, in mmHg) to the fraction of inspired oxygen (FiO₂, expressed as a decimal).
Severity of illness | 27.03.2020-06.05.2024
  Severity of illness during ICU treatment is assessed with validated intensive care unit scores.
Incidence of delirium | 27.03.2020-06.05.2024
  Incidence of delirium in the ICU is measured with validated delirium scores.
Duration of delirium | 27.03.2020-06.05.2024
  Duration of delirium in the ICU is measured in days
Sedation Medications | 27.03.2020-06.05.2024
  Kind of medications required for sedation.
Sedation dosage | 27.03.2020-06.05.2024
  The amount of drug required for sedation.
Duration of sedation | 27.03.2020-06.05.2024
  Duration of sedation is measured in days.
Depth of sedation | 27.03.2020-06.05.2024
  Depth of sedation during ICU treatment
Continuous muscle relaxation | 27.03.2020-06.05.2024
  Continuous muscle relaxation during ICU treatment
Vaccination status | 27.03.2020-06.05.2024
  Vaccination status at the start of ICU treatment
COVID-19-specific immunotherapy | 27.03.2020-06.05.2024
  COVID-19-specific immunotherapy (e.g., tocilizumab, dexamethasone, baricitinib) during ICU treatment
Type of Anti-infective therapy | 27.03.2020-06.05.2024
  Type of anti-infective therapy during ICU treatment
Duration of Anti-infective therapy | 27.03.2020-06.05.2024
  Duration of anti-infective therapy during ICU treatment is measured in days.
Week of pregnancy | 27.03.2020-06.05.2024
  Week of pregnancy during ICU treatment in the pregnant women group
Need for a cesarean section | 27.03.2020-06.05.2024
  Need for a cesarean section in the pregnant women group, yes or no.
Organ complications | 27.03.2020-06.05.2024
  Organ complications, including bleeding and pregnancy complications during hospital treatment. Data from patient records.
Nutrition | 27.03.2020-06.05.2024
  Nutrition (enteral vs. parenteral) during ICU treatment
Dialysis 1 | 27.03.2020-06.05.2024
  Dialysis during ICU treatment (binary)
Dialysis 2 | 27.03.2020-06.05.2024
  Dialysis during ICU treatment (duration)
Intensive care unit mortality | 27.03.2020-06.05.2024
  Data from patient records
Hospital mortality | 27.03.2020-06.05.2024
  Data from patient records
90-day mortality | 27.03.2020-06.05.2024
  Data from patient records
180-day mortality | 27.03.2020-06.05.2024
  Data from patient records
Intensive care unit length of stay | 27.03.2020-06.05.2024
  Participants are followed up for the duration of intensive care unit stay, an expected average of 2 days
Duration of Hospital stay | 27.03.2020-06.05.2024
  Participants are followed up for the duration of hospital stay, an expected average of 7 days
Grip strength Test | 27.03.2020-06.05.2024
  Grip strength at the time of presentation to the PICS outpatient clinic is measured with a dynamometer.
Mobility | 27.03.2020-06.05.2024
  Mobility at the time of presentation to the PICS outpatient clinic is measured with the Timed Up-and-Go (TUG).
Cognition 1 | 27.03.2020-06.05.2024
  Cognition 1 at the time of presentation to the PICS outpatient clinic is measured with the MiniCog. The MiniCog consists of two items, the word recall test and the clock-drawing test. Performance in these test is rated on a scale ranging from 0 - 5, with <3 points indicating a suspicion of dementia.
Cognition 2 | 27.03.2020-06.05.2024
  Cognition 2 at the time of presentation to the PICS outpatient clinic is measured with the Animal Naming Test
Mental health | 27.03.2020-06.05.2024
  Mental health at the time of presentation to the PICS outpatient clinic is measured with Patient Health Questionnaire-4 (It comprises the first two questions of the depression module of the PHQ-D [PHQ-2] and the first two questions of the module for assessing generalized anxiety [GAD-2]) and patient questionnaire with subjective patient assessment.
PBQ Parent-Child Relationship Questionnaire | 27.03.2020-06.05.2024
  PBQ at the time of presentation to the PICS outpatient clinic. This questionnaire is a 25-question self-completion questionnaire, which was developed in order to recognize disorders in the mother-child relationship at an early stage.
  The questionnaire is made up of 4 scales. Scale 1 Delayed attachment cut-off 12, Scale 2 Rejection and anger cut-off 17, Scale 3 Anxiety cut-off 10 and Scale 4 Risk of child abuse cut-off 3.
Edinburgh Postpartum Depression Questionnaire (EPDS) | 27.03.2020-06.05.2024
  The Edinburgh Postnatal Depression Scale (EDPS) was developed to identify women who may have postpartum depression. Each answer is given a score of 0 to 3 .The maximum score is 30. A score of more than 10 suggests minor or major depression may be present.
Health-related quality of life | 27.03.2020-06.05.2024
  Health-related quality of life at the time of presentation to the PICS outpatient clinic is measured with EQ-5D-5L questionnaire. Higher Score indicate better Healt-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany